CLINICAL TRIAL: NCT00788242
Title: The Effect of Glucose-Insulin-Potassium Infusion on Myocardial Injuries and Cardiac Function in Patients Undergoing Cardiac Surgery
Brief Title: The Effect of Glucose-Insulin-Potassium Infusion in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph Ellenberger (Other)
Responsible Party: Sponsor-Investigator, Christoph Ellenberger, Médecin Adjoint, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAC 08-032
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Stenosis; Coronary Heart Disease; Heart Failure
Keywords: Cardiac surgery; Cardioprotection; Aortocoronary bypass graft; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Disease; Heart Failure | interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Administration of glucose-insulin-potassium
  Interventions: Drug: Glucose-insulin-potassium
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucose-insulin-potassium — 20 IU of insulin and 10 mM of KCl mixed with 50 ml of 40% Glucose. Administration of 0.8 ml/kg/h over 60 min before aortic cross-clamping
  Arms: 1
Drug: Placebo — 60 ml of isotonic saline. Administration of 0.8 ml/kg/h over 60 min before aortic cross-clamping
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the cardioprotective effects of a short term infusion of glucose-insulin-potassium (GIK) during heart surgery.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass and ischemic cardiac arrest is associated with a wide spectrum of perioperative myocardial ischemic-reperfusion injuries resulting in significant cardiac morbidity, namely contractile dysfunction, myocardial infarction, and low cardiac output syndrome requiring prolonged intensive care and hospital stay. The infusion of glucose-insulin-potassium (GIK) is one of the oldest cardioprotective interventions during cardiac surgery. Although experimental evidence is strong, clinical data remain conflicting. We will investigate the impact of short term GIK on the extent of myocardial injuries as well as on the left-ventricular systolic and diastolic function in 2 high-risk groups of cardiac surgical patients: Patients with cardiac dysfunction undergoing aortocoronary bypass surgery and patients with severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis
* Coronary artery disease associated with poor left ventricular function
* Parsonnet score >7

Exclusion Criteria:

* Dementia or inability to understand the study protocol
* Off-pump and emergent cardiac surgery
* Poorly controlled diabetes mellitus
* Severe renal insufficiency
* Abnormal liver function Child-Plugh - C
* Body Mass Index < 18 and > 35

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postcardiotomy ventricular dysfunction | 48h postoperative

SECONDARY OUTCOMES:
Systolic and diastolic cardiac function using transoesophageal echocardiography | intraoperative
Hypo-/hyperglycemia Hypo-/hyperkaliemia | intraoperative
Serious cardiovascular adverse events (myocardial infarction, cardiac arrhythmia, low cardiac output, stroke) | 48 postoperative
Serum troponin and creatinine kinase | Intraoperative - 48 h postoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Geneva University Hospital, Geneva, Canton of Geneva
  - Cardiocentro, Lugano, Canton Ticino

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Licker M, Diaper J, Sologashvili T, Ellenberger C. Glucose-insulin-potassium improves left ventricular performances after aortic valve replacement: a secondary analysis of a randomized controlled trial. BMC Anesthesiol. 2019 Sep 6;19(1):175. doi: 10.1186/s12871-019-0845-0. PMID 31492103